CLINICAL TRIAL: NCT04688918
Title: Ultrasound-guided Retrolaminar Block Versus Paravertebral Block for Postoperative Analgesia in Children Undergoing Thoracoscopic Sympathectomy: a Non-inferiority Study
Brief Title: Retrolaminar Block for Pediatric Thoracoscopic Sympathectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Mahmoud Mohammed Alseoudy, Lecturer of anesthesia, ICU & pain management; Faculty of Medicine, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R.20.12.1115
Record Dates: First submitted 2020-12-19; First posted 2020-12-30 (Actual); Last update posted 2023-03-17 (Actual); Status verified 2023-03

CONDITIONS: Pediatric Thoracoscopy

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, double blind study
Who Masked: Participant, Outcomes Assessor
Masking Description: The study subjects and the resident assessing the outcomes will be blinded to the study group. A single investigator will assess the patients for eligibility, obtain written informed consent, open the sealed opaque envelopes containing group allocation
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Retrolamianar block(RLB)) (Active Comparator): Ultrasound-guided RLB with injection of 0.4ml/kglocal anesthestic (bupivacaine) 0.25%will be performed under strict aseptic precautions with ultrasound guidance with patient in the prone position.
  Interventions: Procedure: Retrolaminar block
- Paravertebral group (Active Comparator): Ultrasound-guided paravertebral injection of 0.4ml/kg saline 0.9% will be performed under strict aseptic precautions under ultrasound guidance with patient in the prone position.
  Interventions: Procedure: paravertebral group

INTERVENTIONS:
Procedure: Retrolaminar block — A high-resolution 5-12 MHz linear probe with a sterile cover will be used to perform the block. The patient will be placed in a prone position with a pillow under the chest. The spinous process of the fourth thoracic vertebrae will be identified and marked. Under complete sterilization, the ultrasound high frequency linear probe will be placed in a para-sagittal position, just lateral to the spinous processes of thoracic vertebra, to identify the vertebral lamina. A 50 mm 22-gauge needle will be inserted in an in-plane technique from cranial to caudal direction and will be advanced till hitting the laminae of fourth thoracic vertebrae and then we will try to inject the local anesthetic, if the resistance to injection is very high, hence we will withdraw the needle slowly and its tip will be kept in its position immediately after disappearance this high resistance. Bupivacaine 0.25%, 0.4mL/kg will be injected.
  Arms: Group A (Retrolamianar block(RLB))
Procedure: paravertebral group — A high-resolution 5-12 MHz linear probe with a sterile cover will be used to perform the block. The patient will be placed in a prone position with a pillow under the chest. The transverse process of the fourth thoracic vertebrae will be identified and marked. Under complete sterilization, the ultrasound high frequency linear probe will be placed in a para-sagittal position, just lateral to the spinous processes of thoracic vertebra, to identify the vcostotransverse ligament, 0.4mL/kg will be injected
  Arms: Paravertebral group

SUMMARY:
Thoracoscopic sympathectomy is a rapid and simple technique associated with rare complications, but it is associated with severe postoperative pain that makes breathing and coughing difficult resulting in increased occurrence of pulmonary complications. Paravertebral block has frequently been performed for this procedure but its technical difficulty and safety profile may represent a limitation of its routine use. This prospective, randomized, double-blind controlled study is designed to compare the postoperative analgesic efficacy of ultrasound-guided thoracic retrolaminar block (TRLB) with the paravertebral block in children undergoing thoracoscopic sympathectomy. We hypothesize that ultrasound-guided thoracic retrolaminar block may comparable analgesic effect to paravertebral block with a lesser incidence of complications in pediatric patients undergoing thoracoscopic sympathectomy.

DETAILED DESCRIPTION:
Thoracoscopic sympathectomy is a rapid and simple technique associated with rare complications, but it is associated with severe postoperative pain that makes breathing and coughing difficult resulting in increased occurrence of pulmonary complications, need for analgesic, and hospital stays. Postoperative pain control for pediatric surgeries is a major issue and affects the quality of recovery, parental satisfaction, and surgical success. Opioid usage for pediatric analgesia has many disadvantages, such as postoperative vomiting, pruritus, respiratory depression, and sedation. The introduction of anatomy-based ultrasound (US) imaging for facilitating nerve localization is a major advancement in the field of pediatric regional anesthesia. Paravertebral block has frequently been performed for this procedure but its technical difficulty and safety profile may represent a limitation of its routine use. Ultrasound-guided retrolaminar block (RLB) is a newer alternative to PV block where LA is injected between the lamina and deep paraspinal muscle, rather than between the parietal pleura and costotransverse ligament. This makes it both technically less difficult, but also at less risk of causing substantial side effects such as pneumothorax, inadvertent intrathecal injection, and neurological injury. The analgesic efficacy of RLB has been proven in adults after breast surgery, in patients with multiple rib fractures, and after acute lumbar trauma. This prospective, randomized, double-blind controlled study is designed to compare the postoperative analgesic efficacy of ultrasound-guided thoracic retrolaminar block (TRLB) with the paravertebral block in children undergoing thoracoscopic sympathectomy. We hypothesize that ultrasound-guided thoracic retrolaminar block may comparable analgesic effect to paravertebral block with a lesser incidence of complications in pediatric patients undergoing thoracoscopic sympathectomy. The study will be carried out in Mansoura university children's hospital (MUCH) after obtaining approval from Mansoura Faculty of Medicine Institutional Research Board. Informed written consent will be obtained from the patient guardians'. The planned duration of this study is 8 months. The time gap of the study will be from January 2021 to August 2020.

Eighty children of the American Society of Anesthesiologists physical status I-II of either sex with their age ranging from 8 to 18 years undergoing thoracoscopic surgeries will be recruited for the study.Exclusion criteria will include the history of clinically significant cardiac, hepatic, renal, or neurological dysfunction, coagulopathy, known allergy to amide local anesthetics, and local infection at injection sites.General anesthesia will be induced with incremental sevoflurane in 100% oxygen. After reaching an adequate depth of anesthesia, venous access was established, and then vecuronium will be given in a dose of 0.6 mg/kg and ETT will be inserted. Anesthesia was maintained under controlled ventilation with 1-1.5 MAC of isoflurane and 0.1 mg/kg vecuronium every 30 minutes as a muscle relaxant. Standard intraoperative monitors will be applied for measurement of ECG, heart rate, pulse oximetry, noninvasive blood pressure, and end-tidal carbon dioxide concentration. Baseline readings will be recorded.Computer-generated random numbering of the studied patients will be used for patient randomization before surgery. An opaque sealed envelope will be used and opened in the operative theatre by an anesthesiologist who will not be involved in the current study and who will prepare the drugs used in the study. The anesthesiologist who will be responsible for the patient and the nurse who recorded the patient data will be unaware of the patient's group. Patients will be randomly allocated to one of two equal groups (40 patients for each). Control group (n=40): the patients will receive paravertebral. block.TRLB block group (n=40): ultrasound-guided thoracic retrolaminar block (TRLB).All blocks will be performed by the same anesthetist who is experienced in US-guided pediatric nerve blocks. A high-resolution linear probe with a sterile cover will be used to perform the block. All surgical procedures will be performed by the same surgical team.All blocks will be performed by the same anesthetist who is experienced in US-guided pediatric nerve blocks... All surgical procedures will be performed by the same surgical team.The patient will be placed in a prone position with a pillow under the chest. The spinous process of the fourth thoracic vertebrae will be identified and marked. Under complete sterilization, the ultrasound high-frequency linear probe will be placed in a para-sagittal position, just lateral to the spinous processes of thoracic vertebra, to identify the vertebral lamina. An 80 mm 22-gauge needle will be inserted in an in-plane technique from cranial to the caudal direction and will be advanced till hitting the laminae of the fourth thoracic vertebrae and then we will try to inject the local anesthetic between the lamina and deep paraspinal muscle in RLB group and between the parietal pleura and costotransverse ligament in the paravertebral group. . Bupivacaine 0.25%, 0.4mL/kg will be injected. Vital signs will be recorded every 5 min after the block to ensure the adequacy of the blockade, especially after surgical incision. Surgical procedures will be allowed to start 15 min after the performance of the block. In case of an increase in either patient heart rate to more than 20% of the baseline, fentanyl at 1 ug/kg will be administered. More than 30% decrease in heart rate and systolic blood pressure, respectively, as compared with the baseline values will be treated with atropine or ephedrine as appropriate but the postoperative data of those patients will not be included in the statistical analysis.After completion of the surgery, children will be transferred to the post-anesthesia care unit (PACU) for continuous monitoring of vital signs and for pain assessment. Children will be monitored every 15 min during the first hour in the PACU and every 30 min in the daycare unit until discharge from the hospital. Postoperative analgesia will be measured using vas score 0, 1, 2, 4, 6, 12, 18, 24 hours after surgery. Patients with vas>3 will be given rescue analgesia with 0.05mg/kg morphine intravenously. The primary outcome measure is the total morphine consumption in the first postoperative 24 h. The secondary outcome measures are Postoperative pain score, Time to first rescue analgesia and its frequency, Parent's satisfaction. Block-related complications (pneumothorax, local anesthetic toxicity, or hematoma) and frequency of Nausea and vomiting. Data will be analyzed through SPSS (Statistical Package for Social Sciences). Program version 22. The distribution of data will be first tested by the Shapiro test. Data will be presented as mean and standard deviation (SD), median, and range of numbers and percentages. For normally distributed data, an unpaired t-test will be used to compare between mean values of both groups. For pain score, Mann Whitney U test will be used. Fisher's exact test will be used for comparison of categorical data. The P-value ≤ of 0.05 will be considered as the level of statistical significance.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) status: 1 or 2
* thoracoscopic sympathectomy

Exclusion Criteria

* history of clinically significant cardiac, hepatic, renal, or neurological dysfunction
* coagulopathy
* known allergy to amide local anesthetics
* local infection at injection sites

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-01-03 (Actual); Primary Completion 2023-11-15 (Estimated); Study Completion 2023-12-20 (Estimated)

PRIMARY OUTCOMES:
morphine consumption | Up to 24 hours after the procedure
  The total dose of morphine consumed in first 24 hours will be recorded (mg)

SECONDARY OUTCOMES:
pain score | Up to 24 hours after the procedure
  Pain levels will be assessed post operatively using visual analogue scale(vas),usually 10 centimeters (100 mm) in length, For pain intensity, the scale is most commonly anchored by "no pain" (score of 0) and "pain as bad as it could be" or "worst imaginable pain" (score of 100 [100-mm scale]),vas measured at 0,1, 2, 4, 6, 12, 24 hours
number of patients who will need analgesia | Up to 24 hours after the procedure
  number of patients who request analgesia in the postoperative period
Block related complications | Up to 24 hours after the procedure
  Block related complications (pneumothorax, local anesthetic toxicity or hematoma).[
time of first analgesic request (min) | Up to 24 hours after the procedure
  the time of first analgesic request in first 24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesia, Mansoura University Hospitals, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No